CLINICAL TRIAL: NCT03865134
Title: Evaluation of Visual - Motor Integration and Motor Coordination in Children With Retinopathy of Prematurity
Brief Title: Evaluation of Visual - Motor Development in Children With Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10840098-604.01.01-E.34158
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-02

CONDITIONS: Premature Retinopathy; Visual Impairment; Motor Delay
MeSH Terms: conditions — Retinopathy of Prematurity; Vision Disorders; Psychomotor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laser Group: Children with premature retinopathy treated with Laser therapy. All cases are evaluated with Snellen Test, Autorefractometer, Titmus Stereo Fly Test, Optical Kohlerans Tomography, Peabody Developmental Motor Scales - II. Investigation of Visual Motor Integration will evaluate with Beery- Buktenica Developmental Test of Visual Motor Integration and Peabody. Parents are evaluated World Health Organization Quality of Life - BREF and State - Trait Anxiety Inventory.
  Interventions: Diagnostic Test: Snellen Test; Diagnostic Test: Autorefractometer; Diagnostic Test: Titmus Stereo Fly Test; Diagnostic Test: Optical Kohlerans Tomography; Behavioral: Investigation of Visual Motor Integration; Behavioral: Peabody Developmental Motor Scales - II; Behavioral: World Health Organization Quality of Life - BREF; Behavioral: State - Trait Anxiety Inventory
- Anti-VEGF Group: Children with premature retinopathy treated with anti-VEGF therapy. All cases are evaluated with Snellen Test, Autorefractometer, Titmus Stereo Fly Test, Optical Kohlerans Tomography, Peabody Developmental Motor Scales - II. Investigation of Visual Motor Integration will evaluate with Beery- Buktenica Developmental Test of Visual Motor Integration and Peabody. Parents are evaluated World Health Organization Quality of Life - BREF and State - Trait Anxiety Inventory.
  Interventions: Diagnostic Test: Snellen Test; Diagnostic Test: Autorefractometer; Diagnostic Test: Titmus Stereo Fly Test; Diagnostic Test: Optical Kohlerans Tomography; Behavioral: Investigation of Visual Motor Integration; Behavioral: Peabody Developmental Motor Scales - II; Behavioral: World Health Organization Quality of Life - BREF; Behavioral: State - Trait Anxiety Inventory
- Regrese Group: Children with premature retinopathy haven't applied any invasive treatment method. All cases are evaluated with Snellen Test, Autorefractometer, Titmus Stereo Fly Test, Optical Kohlerans Tomography, Peabody Developmental Motor Scales - II. Investigation of Visual Motor Integration will evaluate with Beery- Buktenica Developmental Test of Visual Motor Integration and Peabody. Parents are evaluated World Health Organization Quality of Life - BREF and State - Trait Anxiety Inventory.
  Interventions: Diagnostic Test: Snellen Test; Diagnostic Test: Autorefractometer; Diagnostic Test: Titmus Stereo Fly Test; Diagnostic Test: Optical Kohlerans Tomography; Behavioral: Investigation of Visual Motor Integration; Behavioral: Peabody Developmental Motor Scales - II; Behavioral: World Health Organization Quality of Life - BREF; Behavioral: State - Trait Anxiety Inventory

INTERVENTIONS:
Diagnostic Test: Snellen Test — Visual acuity measurement
Diagnostic Test: Autorefractometer — Refraction measurement
Diagnostic Test: Titmus Stereo Fly Test — Stereopsis measurement
Diagnostic Test: Optical Kohlerans Tomography — Retinal development measurement
Behavioral: Investigation of Visual Motor Integration — Investigation of visual motor integration, motor coordination and visual perception by Beery- Buktenica Developmental Test of Visual Motor Integration.
Behavioral: Peabody Developmental Motor Scales - II — Evaluation of motor development
Behavioral: World Health Organization Quality of Life - BREF — Assesment of quality of life
Behavioral: State - Trait Anxiety Inventory — Assesment of anxiety

SUMMARY:
The aim of this study was to investigate the eye structure, visual impairment, visual motor development and motor coordination of children between 2-6 ages that had applied to diod laser photocoagulation and intravitreal anti - vascular endothelial growth factor treatment.

DETAILED DESCRIPTION:
There are three different groups in this study. Children between 2-6 ages that had applied to diod laser photocoagulation and intravitreal anti - vascular endothelial growth factor treatment will have evaluated with Snellen Test, Titmus Fly Test, Optical Kohlerans Tomography, Beery-Buktenica Developmental Test of Visual Motor Integration, Peabody Developmental Motor Scales-II, World Health Organization Quality of Life - BREF and State - Trait Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 2-6 years of age
* Gestational age range 26-34. be between weeks
* To be diagnosed with retinopathy of prematurity
* Neurological, hereditary and not having metabolic disease
* Compliance with visual examinations and physiotherapy evaluations
* To be children and parents who agree to participate in the study

Exclusion Criteria:

* To be a child who does not comply with Optical Kohlerans Tomography (OCT)
* Not participating in one or more of the eye examination or physiotherapy assessments
* Being children and parents who do not agree to participate in the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants who were followed up and treated in the outpatient clinic of Zeynep Kamil Women and Children Diseases Training and Research Hospital, Ophthalmology Clinic with the diagnosis of Prematurity Retinopathy between the years 2012-2015 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Visual Motor Integration | 3 weeks
  Visual-motor integration (VMI) is "the degree to which visual perception and finger-hand movements are well coordinated" and will asses with Beery-Buktenica Developmental Test of Visual-Motor Integration in this study. This test is a standardized, norm-referenced assessment involving copying geometric forms that is used to determine the level of integration between visual and motor systems in people of all ages.
  The Short Format and Full Format tests take about 10-15 minutes each to administer. Results are reported as standard scores, percentiles, and age equivalents.
Visual Perception | 3 weeks
  Visual perception will asses with Beery-Buktenica Developmental Test of Visual-Motor Integration in this study. This test is a standardized, norm-referenced assessment involving copying geometric forms that is used to determine the level of integration between visual and motor systems in people of all ages. Visual Perception test takes about 5 minutes. Results are reported as standard scores, percentiles, and age equivalents.
Motor Coordination | 3 weeks
  Motor Coordination is coordination of finger movements and will asses by Beery-Buktenica Developmental Test of Visual-Motor Integration in this study. This test is a standardized, norm-referenced assessment involving copying geometric forms that is used to determine the level of integration between visual and motor systems in people of all ages. Motor coordination test takes about 5 minutes. Results are reported as standard scores, percentiles, and age equivalents.
Retinal Layers' Development | 3 weeks
  Development of retinal layers will assess with Optical coherence tomography (OCT). The OCT allows for in vivo, cross-sectional assessment of eye tissue, including the retina and its vasculature. By comparing the interference patterns of light that passes through live tissue to a reference arm, OCT provides high-resolution imaging of just a few microns of eye microanatomy.

OTHER OUTCOMES:
Quality of Life in Parents | 3 weeks
  Quality of life assessment of parents will evaluate with The WHOQOL-BREF instrument that is comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.
State - Trait Anxiety of Parents | 3 weeks
  State and trait anxiety level of parents will asses by the State-Trait Anxiety Inventory (STAI) that is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress.The STAI has 20 items for assessing trait anxiety and 20 for state anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Candan Algun, Study Director — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rothman AL, Mangalesh S, Chen X, Toth CA. Optical coherence tomography of the preterm eye: from retinopathy of prematurity to brain development. Eye Brain. 2016 May 27;8:123-133. doi: 10.2147/EB.S97660. eCollection 2016. PMID 28539807
- [Background] Kabatas EU, Kurtul BE, Altiaylik Ozer P, Kabatas N. Comparison of Intravitreal Bevacizumab, Intravitreal Ranibizumab and Laser Photocoagulation for Treatment of Type 1 Retinopathy of Prematurity in Turkish Preterm Children. Curr Eye Res. 2017 Jul;42(7):1054-1058. doi: 10.1080/02713683.2016.1264607. Epub 2017 Jan 27. PMID 28128986
- [Result] Araz-Ersan B, Kir N, Tuncer S, Aydinoglu-Candan O, Yildiz-Inec D, Akdogan B, Ekici B, Demirel A, Ozmen M. Preliminary anatomical and neurodevelopmental outcomes of intravitreal bevacizumab as adjunctive treatment for retinopathy of prematurity. Curr Eye Res. 2015 May;40(6):585-91. doi: 10.3109/02713683.2014.941070. Epub 2014 Jul 15. PMID 25025864